CLINICAL TRIAL: NCT00805051
Title: Does an Acquired Von Willebrand Syndrome Influence Perioperative Blood Loss in Patients With Severe Aortic Stenosis Undergoing Aortic Valve Replacement?
Brief Title: Acquired Von Willebrand Syndrome in Severe Aortic Stenosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Daniel Bolliger, PD Dr. Daniel Bolliger, University Hospital, Basel, Switzerland
Other Study IDs: 07/08
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Bleeding; Von Willebrand Disease; Aortic Stenosis
Keywords: Aortic stenosis; aortic valve replacement; von Willebrand disease; blood loss
MeSH Terms: conditions — Hemorrhage; von Willebrand Diseases; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe aortic stenosis: Patients undergoing aortic valve replacement because of severe aortic stenosis

SUMMARY:
Patients with severe aortic stenosis often suffer from an acquired Von Willebrand syndrome by degeneration of the polymers during passage through the narrow valve leading to turbulences. We hypothesized that the diagnosis of acquired von Willebrand syndrome influence perioperative blood loss in patients undergoing open cardiac valve replacement.

DETAILED DESCRIPTION:
Patients with severe aortic stenosis often suffer from an acquired Von Willebrand syndrome by degeneration of the polymers during passage through the narrow valve leading to turbulences. After written consent and an extended anamnesis of existing coagulopathy, we take three blood samples in these patients: before surgery, on the day after surgery and 4 weeks after surgery. We determine von Willebrand factor in lab and by a point-of-care platelet function analyzer (Multiplate TM). We measure amount of mediastinal drainage after 24 hours and blood product consumption in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis (Orifice area < 1 cm2)

Exclusion Criteria:

* missing consent
* severe hepatic or renal disfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for aortic valve replacement for severe aortic stenosis
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Amount of mediastinal drainage in the first 24 hours | 24 hours

SECONDARY OUTCOMES:
Amount of given blood products in the first 24 hours | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Miodrag Filipovic, MD, Principal Investigator — Department of Anaesthesia, University of Basel Hospital
Locations (1):
- Department of Anaesthesia, University of Basel Hospital, Basel, Switzerland